CLINICAL TRIAL: NCT04796844
Title: Mild/Moderate Asthma Network of Italy Observatory
Brief Title: MANI Real-life Perspective Observatory
Acronym: MANI
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Pneumologia (Other)
Collaborators: Società Italiana di Allergologia, Asma e Immunologia Clinica (Other)
Responsible Party: Sponsor
Other Study IDs: 456/2020 - DB id 10481; MANI Project (Other: SIP/IRS and SIAAIC)
Record Dates: First submitted 2021-02-23; First posted 2021-03-15 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Asthma; Mild Asthma; Moderate Asthma
Keywords: Asthma; Adult; Cluster; Cohort study; Italy; Prospective
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The information collected in the CRF coincides with the patient data routinely reported in the medical record.
  In case of a blood draw for routine clinical practice, a blood sample will be acquired and stored to assess biomarkers currently under investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry aims is to collect a large number of patients with mild and moderate asthma in a real-word conditions for a perspective observation of epidemiological evolution of the disease in relation to the therapeutic interventions available currently and in the near future.

DETAILED DESCRIPTION:
To represent real-world mild moderate Italian asthmatics, all adults with diagnosed asthma by specialist, according GINA (Global Initiative for Asthma) document, attending respiratory or allergy clinic for a scheduled visit are eligible for study enrollment. If inclusion/exclusion criteria are satisfied, a written consent to participate in the study will be obtained and an informative leaflet for the patient and his/her general practitioners will be delivered.

Subjects follow up will be scheduled according with GINA document and center plan (6 or 12 months follow up visit).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Asthma diagnosis according GINA 2020 algorithm (Annex 1)
* Patients enrolled in other previous or ongoing observational studies

Exclusion Criteria:

* Severe asthma patients according International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. [Chung KF et al. European Respiratory Journal Feb 2014, 43 (2) 343-373; DOI: 10.1183/09031936.00202013 (Annex 2)]
* Subjects are excluded from this cohort if they exhibit interstitial lung diseases, pulmonary neoplasms, current lung infections, immunological disorders leading to the use of immunosuppressants or continuous treatment with oral steroids.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To represent real-world mild moderate Italian asthmatics, all adults with diagnosed asthma by specialist, according GINA document, attending respiratory or allergy clinic for a scheduled visit are eligible for study enrollment. If inclusion/exclusion criteria are satisfied, a written consent to participate in the study will be obtained and an informative leaflet for the patient and his/her GPs will be delivered.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
A cluster-based, real world, cross-sectional perspective, observational cohort study | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Perspective observation of epidemiological evolution of mild and moderate asthma (rate of asthmatic patients transitioned to a more severe stage according Global Initiative for Asthma [GINA] document)

SECONDARY OUTCOMES:
Real life assessment of control, exacerbation and PROs in patients treated with different drugs and schedule | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Real-life assessment of asthma control over time (Asthma Control Test and Asthma Control Questionnaire scores), exacerbation rate over time (n/year) and patient-reported outcomes (e.g., quality of life, patient engagement, disease awareness) from groups treated with different drugs and schedules (questionnaire score)
Asthma control in pregnant women | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Asthma control in pregnant women by means of a specific application for android- and iOS-based smartphones, in comparison with the traditional current management
Burden of OCS in mild and moderate asthma | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Burden of oral corticosteroids in mild and moderate asthma (mg/year)
SABA use in mild and moderate asthma | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  SABA use in mild and moderate asthma (canisters/year)
Influence of infections and vaccinations on disease outcomes and progression | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Influence of infections and vaccinations on disease outcomes and progression (rate of progression; questionnaire score)
Influence of upper airway disease on disease outcomes and progression | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Influence of upper airway disease on disease outcomes and progression (rate of progression; questionnaire score)
Impact of inhalation techniques and smart inhalers on disease outcomes and progression | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Impact of inhalation techniques and smart inhalers on disease outcomes and progression (inhalation error/asthma control score; inhalation error/rate of progression)
Environmental exposure influences on disease outcome and progression | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Environmental exposure influences on disease outcome and progression (PM10/rate of progression)
Evolution of inflammatory patterns over time | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Evolution of inflammatory patterns over time and their relationships to disease outcomes and progression (published biomarker value/asthma control; published biomarker value/rate of progression)
Role of smoking and life style in lung function and disease progression | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Role of smoking and life style in lung function and disease progression (pack year/disease progression)
Patients reported outcomes over time | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Patients reported outcomes over time (score according validated questionnaires)
Patient awareness and engagement in mild and moderate asthma | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Patient awareness and engagement in mild and moderate asthma (questionnaire score)
Impact of digital therapy on disease management and outcomes | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Impact of digital therapy on disease management and outcomes (canister/year and dose/year)
Direct, indirect, and intangible costs of mild and moderate asthma | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Direct, indirect, and intangible costs of mild and moderate asthma (EU/disease severity)
Cost-efficiency of mild/moderate asthma treatments and management plans | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Cost-efficiency of mild/moderate asthma treatments and management plans (cost/year)
Sociodemographic issues related to disease progression and burden | through study completion; follow-up procedures will last 10 years from the date of the last patient enrolled
  Sociodemographic issues related to disease progression and burden (age, sex, education, employment/rate of progression)

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Braido, Principal Investigator — IRCCS Ospedale Policlinico San Martino, Department of Internal Medicine (DiMI), University of Genoa
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, Italy

REFERENCES:
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Derived] Braido F, Blasi F, Canonica GW, Paggiaro P, Beghe B, Bonini M, Carpagnano GE, Del Giacco S, Lavorini F, Milanese M, Patella V, Santus P, Contoli M; MANI Network; Allegrini C, Baiardini I, Bonzano L, Caiaffa MF, Castelnuovo P, Corsico AG, Cosmi L, Costantino MT, Cottini M, Crimi N, Crivellaro MA, D'Alo S, Folletti I, Fornari D, Foschino-Barbaro MP, Franceschini L, Gargano D, Oliani KL, Maniscalco M, Melissari L, Montagni M, Montuschi P, Murgia N, Pannofino A, Papi A, Parente R, Pelaia G, Pini L, Puggioni F, Pulera N, Resta O, Ricciardi L, Ridolo E, Savi E, Savoia F, Scala G, Senna G, Tripodi S, Vatrella A, Ventura MT, Viviano VM, Yacoub MR. Mild/Moderate Asthma Network in Italy (MANI): a long-term observational study. J Asthma. 2022 Sep;59(9):1908-1913. doi: 10.1080/02770903.2021.1968895. Epub 2021 Sep 1. PMID 34469268

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04796844/Prot_SAP_000.pdf